CLINICAL TRIAL: NCT03082976
Title: PREDICT: Prevalence of BRCA1 and BRCA2 Mutations in Ovarian Cancer Patients in the Gulf Region. A Prospective, Multi-centre, Epidemiological Observational Study Designed to Evaluate the Prevalence of BRCA1 and BRCA2 Mutations in Current and Newly Diagnosed Ovarian Cancer Patients Across Different Countries in the Gulf Region. This Study Study Will Also Describe the Epidemiological Features for the Disease for the Enrolled Patients.
Brief Title: Prevalence of BRCA1 and BRCA2 Mutations in Ovarian Cancer Patients in the Gulf Region
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00118
Record Dates: First submitted 2017-02-27; First posted 2017-03-17 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, multi-centre, epidemiological observational study designed to evaluate the prevalence of BRCA1 and BRCA2 (BReast CAncer gene) mutations in current and newly diagnosed ovarian cancer patients across different countries in the Gulf region. This study will also describe the epidemiological features for the disease for the enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing to sign the informed consent form (ICF)
2. Female subjects 18 years of age or older
3. Have histologically confirmed diagnosis of Federation of Gynecology and Obstetrics (FIGO) ovarian epithelial, primary peritoneal cancer made by one or more of the following:

   1. Standard staging laparotomy including bilateral salpingo-oophorectomy,omentectomy, and lymph node sampling and debulking and/or
   2. Surgical resection and radiographic evidence consistent with ovarian cancer
   3. Paracentesis or biopsy with radiographic evidence consistent with ovarian cancer(normal appearing pancreas, liver, and gastrointestinal tract).
4. Have availability of paraffin-embedded archived tumor tissue block (preferred) or, if a block is not possible, a minimum of twenty 10-um sections.

Exclusion Criteria:

Patients who meet any of the following criteria are ineligible to participate in the study and hence will not be consented:

1. The diagnosis is not of a primary ovarian cancer; thus, patients will be excluded if a previous cancer has metastasized to the ovary, or if there is a secondary malignancy that is associated with the ovarian cancer.
2. Is not able or willing to provide written informed consent.
3. Have a diagnosis of other severe acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of the study.
4. Be a patient who, in the judgment of the Investigator, would be inappropriate for enrollment in this study.

A rationale will be documented for all patients who are screened and ultimately excluded from the study as a result of meeting any of the aforementioned exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will be women at least 18 years of age with histologically confirmed ovarian, peritoneal, and fallopian tube cancers at participating oncology hospitals/departments in the Gulf region. Patients enrolled in this study will be assigned to either the treatment-experienced subgroup for those who were previously diagnosis and are undergoing treatment at the time of enrollment, or the treatment-native group for those who were recently diagnosed and not yet undergoing treatment.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Prevalence of somatic BRCA mutations among ovarian cancer patients | Up to 4 Weeks for BRCA testing result
  The primary objective of this study is to discern the prevalence of somatic BRCA1 and BRCA2 mutations in patients with ovarian cancer, peritoneal cancer, and fallopian tube cancer, as assessed by tissue genetic testing in tumor samples

SECONDARY OUTCOMES:
Associations or correspondence in prevalence between genetic alterations | Up to 4 Weeks for BRCA testing result
  Examine associations (or correspondence) in prevalence between genetic alterations in hereditary (germline) and tissue (somatic) BRCA mutations by testing for germline (blood) mutations in those patients who are known to have somatic mutations
Describe epidemiological characteristics | Up to 4 Weeks for BRCA testing result
  Describe epidemiological characteristics (e.g., age, ethnicities) of patients being treated for ovarian cancer.
Describe treatment modalities | Up to 4 Weeks for BRCA testing result
  Describe treatment strategy among the treatment-experienced subgroup of patients who were previously diagnosed with ovarian cancer
Categorize epideimiological charactersitics and clinical features | Up to 4 Weeks for BRCA testing result
  Describe epidemiological characteristics(e.g. Comorbidities, stage) of patients being treated for ovarian cancer

OTHER OUTCOMES:
Compare standards of care practices | Up to 4 Weeks for BRCA testing result
  An exploratory objective is to compare standards of care and pre- and post-diagnosis practices in each country, for example, with respect to tissue collection, processing, storage and maintenance, which is of great importance to future studies building on the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Jaloudi, MD, Principal Investigator — Tawam Hospital
Locations (1):
- Research Site, Al Ain City, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azribi F, Abdou E, Dawoud E, Ashour M, Kamal A, Al Sayed M, Burney I. Prevalence of BRCA1 and BRCA2 pathogenic sequence variants in ovarian cancer patients in the Gulf region: the PREDICT study. BMC Cancer. 2021 Dec 20;21(1):1350. doi: 10.1186/s12885-021-09094-8. PMID 34930165
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00118&attachmentIdentifier=8c8c54f3-fe1d-475e-827e-76cf519cf918&fileName=CSR_PREDICT_V4.D133FR00118redacted.pdf&versionIdentifier=